CLINICAL TRIAL: NCT02490124
Title: The Effect of Type 1 Diabetes on Pan-Arterial Vascular Function and Insulin Sensitivity in Humans
Acronym: EJB046
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Eugene Barrett, Professor Eugene Barrett MD PhD, University of Virginia
Other Study IDs: 17099
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Type 1
Keywords: Diabetes Type 1; Vascular Function
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetic: Type 1 Diabetic
- Control: normal healthy control

SUMMARY:
Arterial vascular disease is the major cause of morbidity and mortality for Type 1 diabetic patients (DM1). Metabolic insulin resistance (metIR), even in the absence of hyperglycemia, conveys a 1.5 to 3-fold increased CVD risk in the general population. Metabolic Insulin Resistance (MetIR) has been repeatedly shown to be prevalent in adults and adolescents with DM1. MetIR in obesity and DM2 are accompanied by vascular insulin resistance (vasIR) which is characterized by impaired vasodilatory action of insulin on resistance or microvascular vessels. VasIR has not been systematically studied in DM1. We hypothesize that in young adults DM1 impairs both baseline and insulin-responsive vascular function throughout the arterial vasculature.

DETAILED DESCRIPTION:
In our study, 20 healthy control subjects will be compared to 20 DM1 patients (18-40 yrs). We will assess function in conduit (pulse wave velocity-PWV, flow-mediated dilation-FMD and augmentation index-AI), resistance (post-ischemic flow velocity-PIFV) and heart and skeletal muscle microvascular (contrast enhanced ultrasound-CEU) vessels before and after 2 hrs of a euglycemic insulin clamp.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* BMI ≤ 25
* Healthy with no chronic illness (control group only)
* Normal screening labs or no clinically significant values
* DM1 subjects will have been on insulin for at least 5 years and HbA1c <9

Exclusion Criteria:

* First degree relative with Type 1 or 2 Diabetes (for control group only)
* Smoking presently or in the past 6 months
* Medications that affect the vasculature (except ACE or ARB in DM1 subjects, although they will need to be off these drugs for 2 weeks prior to study).
* Elevated LDL cholesterol > 160
* BP <100/60 or >160/90
* Pulse oximetry <90%
* Pregnant or breastfeeding
* History of cardiovascular disease, cerebral vascular disease, peripheral vascular disease, liver disease
* Presence of an intracardiac or intrapulmonary shunt (we will screen for this by auscultation during the physical exam ).
* Known hypersensitivity to perflutren (contained in Definity)
* For DM1 group:

  * HbA1c ≥ 9
  * Microalbuminuria
  * Retinipathy
  * Ketoacidosis within the past year.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Type 1 Diabetes Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Augmentation Index | baseline
  vascular measure
Pulse Wave Velocity | baseline
  vascular measure
Flow Mediated Dilation | Baseline
  vascular measure
Contrast Enhanced Ultrasound | baseline
  vascular measure
Augmentation Index | after 2 hour insulin clamp
  vascular measure
Pulse Wave Velocity | after 2 hour insulin clamp
  vascular measure
Flow Mediated Dilation | after 2 hour insulin clamp
  vascular measure
Contrast Enhanced Ultrasound | after 2 hour insulin clamp
  vascular measure

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J. B, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Libby P, Nathan DM, Abraham K, Brunzell JD, Fradkin JE, Haffner SM, Hsueh W, Rewers M, Roberts BT, Savage PJ, Skarlatos S, Wassef M, Rabadan-Diehl C; National Heart, Lung, and Blood Institute; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Report of the National Heart, Lung, and Blood Institute-National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Circulation. 2005 Jun 28;111(25):3489-93. doi: 10.1161/CIRCULATIONAHA.104.529651. No abstract available. PMID 15983263
- [Background] Krolewski AS, Kosinski EJ, Warram JH, Leland OS, Busick EJ, Asmal AC, Rand LI, Christlieb AR, Bradley RF, Kahn CR. Magnitude and determinants of coronary artery disease in juvenile-onset, insulin-dependent diabetes mellitus. Am J Cardiol. 1987 Apr 1;59(8):750-5. doi: 10.1016/0002-9149(87)91086-1. PMID 3825934
- [Background] Widlansky ME, Gokce N, Keaney JF Jr, Vita JA. The clinical implications of endothelial dysfunction. J Am Coll Cardiol. 2003 Oct 1;42(7):1149-60. doi: 10.1016/s0735-1097(03)00994-x. PMID 14522472
- [Background] Schram MT, Chaturvedi N, Schalkwijk CG, Fuller JH, Stehouwer CD; EURODIAB Prospective Complications Study Group. Markers of inflammation are cross-sectionally associated with microvascular complications and cardiovascular disease in type 1 diabetes--the EURODIAB Prospective Complications Study. Diabetologia. 2005 Feb;48(2):370-8. doi: 10.1007/s00125-004-1628-8. Epub 2005 Feb 4. PMID 15692810
- [Background] Johnstone MT, Creager SJ, Scales KM, Cusco JA, Lee BK, Creager MA. Impaired endothelium-dependent vasodilation in patients with insulin-dependent diabetes mellitus. Circulation. 1993 Dec;88(6):2510-6. doi: 10.1161/01.cir.88.6.2510. PMID 8080489
- [Background] Clarkson P, Celermajer DS, Donald AE, Sampson M, Sorensen KE, Adams M, Yue DK, Betteridge DJ, Deanfield JE. Impaired vascular reactivity in insulin-dependent diabetes mellitus is related to disease duration and low density lipoprotein cholesterol levels. J Am Coll Cardiol. 1996 Sep;28(3):573-9. doi: 10.1016/0735-1097(96)82380-1. PMID 8772741
- [Background] Lockhart CJ, Agnew CE, McCann A, Hamilton PK, Quinn CE, McCall DO, Plumb RD, McClenaghan VC, McGivern RC, Harbinson MT, McVeigh GE. Impaired flow-mediated dilatation response in uncomplicated Type 1 diabetes mellitus: influence of shear stress and microvascular reactivity. Clin Sci (Lond). 2011 Aug;121(3):129-39. doi: 10.1042/CS20100448. PMID 21345174
- [Background] Boutouyrie P, Tropeano AI, Asmar R, Gautier I, Benetos A, Lacolley P, Laurent S. Aortic stiffness is an independent predictor of primary coronary events in hypertensive patients: a longitudinal study. Hypertension. 2002 Jan;39(1):10-5. doi: 10.1161/hy0102.099031. PMID 11799071
- [Background] Anderson TJ, Charbonneau F, Title LM, Buithieu J, Rose MS, Conradson H, Hildebrand K, Fung M, Verma S, Lonn EM. Microvascular function predicts cardiovascular events in primary prevention: long-term results from the Firefighters and Their Endothelium (FATE) study. Circulation. 2011 Jan 18;123(2):163-9. doi: 10.1161/CIRCULATIONAHA.110.953653. Epub 2011 Jan 3. PMID 21200002
- [Background] Schauer IE, Snell-Bergeon JK, Bergman BC, Maahs DM, Kretowski A, Eckel RH, Rewers M. Insulin resistance, defective insulin-mediated fatty acid suppression, and coronary artery calcification in subjects with and without type 1 diabetes: The CACTI study. Diabetes. 2011 Jan;60(1):306-14. doi: 10.2337/db10-0328. Epub 2010 Oct 26. PMID 20978091
- [Background] Liu J, Jahn LA, Fowler DE, Barrett EJ, Cao W, Liu Z. Free fatty acids induce insulin resistance in both cardiac and skeletal muscle microvasculature in humans. J Clin Endocrinol Metab. 2011 Feb;96(2):438-46. doi: 10.1210/jc.2010-1174. Epub 2010 Nov 3. PMID 21047922
- [Background] Laakso M, Edelman SV, Brechtel G, Baron AD. Decreased effect of insulin to stimulate skeletal muscle blood flow in obese man. A novel mechanism for insulin resistance. J Clin Invest. 1990 Jun;85(6):1844-52. doi: 10.1172/JCI114644. PMID 2189893
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Verma S, Buchanan MR, Anderson TJ. Endothelial function testing as a biomarker of vascular disease. Circulation. 2003 Oct 28;108(17):2054-9. doi: 10.1161/01.CIR.0000089191.72957.ED. No abstract available. PMID 14581384
- [Background] Barrett EJ, Wang H, Upchurch CT, Liu Z. Insulin regulates its own delivery to skeletal muscle by feed-forward actions on the vasculature. Am J Physiol Endocrinol Metab. 2011 Aug;301(2):E252-63. doi: 10.1152/ajpendo.00186.2011. Epub 2011 May 24. PMID 21610226
- [Background] Keske MA, Clerk LH, Price WJ, Jahn LA, Barrett EJ. Obesity blunts microvascular recruitment in human forearm muscle after a mixed meal. Diabetes Care. 2009 Sep;32(9):1672-7. doi: 10.2337/dc09-0206. Epub 2009 Jun 1. PMID 19487636
- [Background] Miyaki A, Maeda S, Yoshizawa M, Misono M, Saito Y, Sasai H, Endo T, Nakata Y, Tanaka K, Ajisaka R. Effect of weight reduction with dietary intervention on arterial distensibility and endothelial function in obese men. Angiology. 2009 Jun-Jul;60(3):351-7. doi: 10.1177/0003319708325449. Epub 2008 Nov 19. PMID 19022788
- [Background] Sugawara J, Otsuki T, Tanabe T, Hayashi K, Maeda S, Matsuda M. Physical activity duration, intensity, and arterial stiffening in postmenopausal women. Am J Hypertens. 2006 Oct;19(10):1032-6. doi: 10.1016/j.amjhyper.2006.03.008. PMID 17027823
- [Background] Baron AD, Steinberg HO, Chaker H, Leaming R, Johnson A, Brechtel G. Insulin-mediated skeletal muscle vasodilation contributes to both insulin sensitivity and responsiveness in lean humans. J Clin Invest. 1995 Aug;96(2):786-92. doi: 10.1172/JCI118124. PMID 7635973
- [Background] Barrett EJ, Eggleston EM, Inyard AC, Wang H, Li G, Chai W, Liu Z. The vascular actions of insulin control its delivery to muscle and regulate the rate-limiting step in skeletal muscle insulin action. Diabetologia. 2009 May;52(5):752-64. doi: 10.1007/s00125-009-1313-z. Epub 2009 Mar 13. PMID 19283361
- [Background] Pearson TA, Mensah GA, Alexander RW, Anderson JL, Cannon RO 3rd, Criqui M, Fadl YY, Fortmann SP, Hong Y, Myers GL, Rifai N, Smith SC Jr, Taubert K, Tracy RP, Vinicor F; Centers for Disease Control and Prevention; American Heart Association. Markers of inflammation and cardiovascular disease: application to clinical and public health practice: A statement for healthcare professionals from the Centers for Disease Control and Prevention and the American Heart Association. Circulation. 2003 Jan 28;107(3):499-511. doi: 10.1161/01.cir.0000052939.59093.45. No abstract available. PMID 12551878
- [Background] Schalkwijk CG, Poland DC, van Dijk W, Kok A, Emeis JJ, Drager AM, Doni A, van Hinsbergh VW, Stehouwer CD. Plasma concentration of C-reactive protein is increased in type I diabetic patients without clinical macroangiopathy and correlates with markers of endothelial dysfunction: evidence for chronic inflammation. Diabetologia. 1999 Mar;42(3):351-7. doi: 10.1007/s001250051162. PMID 10096789
- [Background] Ladeia AM, Stefanelli E, Ladeia-Frota C, Moreira A, Hiltner A, Adan L. Association between elevated serum C-reactive protein and triglyceride levels in young subjects with type 1 diabetes. Diabetes Care. 2006 Feb;29(2):424-6. doi: 10.2337/diacare.29.02.06.dc05-2033. No abstract available. PMID 16443901
- [Background] Sundell J, Ronnemaa T, Laine H, Raitakari OT, Luotolahti M, Nuutila P, Knuuti J. High-sensitivity C-reactive protein and impaired coronary vasoreactivity in young men with uncomplicated type 1 diabetes. Diabetologia. 2004 Nov;47(11):1888-94. doi: 10.1007/s00125-004-1543-z. Epub 2004 Nov 24. PMID 15565375
- [Background] Hayaishi-Okano R, Yamasaki Y, Katakami N, Ohtoshi K, Gorogawa S, Kuroda A, Matsuhisa M, Kosugi K, Nishikawa N, Kajimoto Y, Hori M. Elevated C-reactive protein associates with early-stage carotid atherosclerosis in young subjects with type 1 diabetes. Diabetes Care. 2002 Aug;25(8):1432-8. doi: 10.2337/diacare.25.8.1432. PMID 12145246
- [Background] Nagaoka T, Kuo L, Ren Y, Yoshida A, Hein TW. C-reactive protein inhibits endothelium-dependent nitric oxide-mediated dilation of retinal arterioles via enhanced superoxide production. Invest Ophthalmol Vis Sci. 2008 May;49(5):2053-60. doi: 10.1167/iovs.07-1387. PMID 18436840
- [Background] Qamirani E, Ren Y, Kuo L, Hein TW. C-reactive protein inhibits endothelium-dependent NO-mediated dilation in coronary arterioles by activating p38 kinase and NAD(P)H oxidase. Arterioscler Thromb Vasc Biol. 2005 May;25(5):995-1001. doi: 10.1161/01.ATV.0000159890.10526.1e. Epub 2005 Feb 17. PMID 15718491
- [Background] Colhoun HM, Betteridge DJ, Durrington PN, Hitman GA, Neil HA, Livingstone SJ, Thomason MJ, Mackness MI, Charlton-Menys V, Fuller JH; CARDS investigators. Primary prevention of cardiovascular disease with atorvastatin in type 2 diabetes in the Collaborative Atorvastatin Diabetes Study (CARDS): multicentre randomised placebo-controlled trial. Lancet. 2004 Aug 21-27;364(9435):685-96. doi: 10.1016/S0140-6736(04)16895-5. PMID 15325833
- [Background] Behrendt D, Ganz P. Endothelial function. From vascular biology to clinical applications. Am J Cardiol. 2002 Nov 21;90(10C):40L-48L. doi: 10.1016/s0002-9149(02)02963-6. PMID 12459427
- [Background] Szmitko PE, Wang CH, Weisel RD, de Almeida JR, Anderson TJ, Verma S. New markers of inflammation and endothelial cell activation: Part I. Circulation. 2003 Oct 21;108(16):1917-23. doi: 10.1161/01.CIR.0000089190.95415.9F. No abstract available. PMID 14568885
- [Background] de Graaf JC, Banga JD, Moncada S, Palmer RM, de Groot PG, Sixma JJ. Nitric oxide functions as an inhibitor of platelet adhesion under flow conditions. Circulation. 1992 Jun;85(6):2284-90. doi: 10.1161/01.cir.85.6.2284. PMID 1591842
- [Background] Joannides R, Haefeli WE, Linder L, Richard V, Bakkali EH, Thuillez C, Luscher TF. Nitric oxide is responsible for flow-dependent dilatation of human peripheral conduit arteries in vivo. Circulation. 1995 Mar 1;91(5):1314-9. doi: 10.1161/01.cir.91.5.1314. PMID 7867167
- [Background] Esteve E, Castro A, Lopez-Bermejo A, Vendrell J, Ricart W, Fernandez-Real JM. Serum interleukin-6 correlates with endothelial dysfunction in healthy men independently of insulin sensitivity. Diabetes Care. 2007 Apr;30(4):939-45. doi: 10.2337/dc06-1793. PMID 17392554
- [Background] Clausen P, Jacobsen P, Rossing K, Jensen JS, Parving HH, Feldt-Rasmussen B. Plasma concentrations of VCAM-1 and ICAM-1 are elevated in patients with Type 1 diabetes mellitus with microalbuminuria and overt nephropathy. Diabet Med. 2000 Sep;17(9):644-9. doi: 10.1046/j.1464-5491.2000.00347.x. PMID 11051283
- [Background] Moncada S, Higgs A. The L-arginine-nitric oxide pathway. N Engl J Med. 1993 Dec 30;329(27):2002-12. doi: 10.1056/NEJM199312303292706. No abstract available. PMID 7504210
- [Background] Steinberg HO, Brechtel G, Johnson A, Fineberg N, Baron AD. Insulin-mediated skeletal muscle vasodilation is nitric oxide dependent. A novel action of insulin to increase nitric oxide release. J Clin Invest. 1994 Sep;94(3):1172-9. doi: 10.1172/JCI117433. PMID 8083357
- [Background] Steinberg HO, Chaker H, Leaming R, Johnson A, Brechtel G, Baron AD. Obesity/insulin resistance is associated with endothelial dysfunction. Implications for the syndrome of insulin resistance. J Clin Invest. 1996 Jun 1;97(11):2601-10. doi: 10.1172/JCI118709. PMID 8647954
- [Background] Rossi R, Cioni E, Nuzzo A, Origliani G, Modena MG. Endothelial-dependent vasodilation and incidence of type 2 diabetes in a population of healthy postmenopausal women. Diabetes Care. 2005 Mar;28(3):702-7. doi: 10.2337/diacare.28.3.702. PMID 15735211
- [Background] Vincent MA, Barrett EJ, Lindner JR, Clark MG, Rattigan S. Inhibiting NOS blocks microvascular recruitment and blunts muscle glucose uptake in response to insulin. Am J Physiol Endocrinol Metab. 2003 Jul;285(1):E123-9. doi: 10.1152/ajpendo.00021.2003. PMID 12791603
- [Background] Eggleston EM, Jahn LA, Barrett EJ. Hyperinsulinemia rapidly increases human muscle microvascular perfusion but fails to increase muscle insulin clearance: evidence that a saturable process mediates muscle insulin uptake. Diabetes. 2007 Dec;56(12):2958-63. doi: 10.2337/db07-0670. Epub 2007 Aug 24. PMID 17720897
- [Background] Rattigan S, Clark MG, Barrett EJ. Acute vasoconstriction-induced insulin resistance in rat muscle in vivo. Diabetes. 1999 Mar;48(3):564-9. doi: 10.2337/diabetes.48.3.564. PMID 10078557
- [Background] Clark AD, Barrett EJ, Rattigan S, Wallis MG, Clark MG. Insulin stimulates laser Doppler signal by rat muscle in vivo, consistent with nutritive flow recruitment. Clin Sci (Lond). 2001 Mar;100(3):283-90. PMID 11222114
- [Background] Llaurado G, Simo R, Villaplana M, Berlanga E, Vendrell J, Gonzalez-Clemente JM. Can augmentation index substitute aortic pulse wave velocity in the assessment of central arterial stiffness in type 1 diabetes? Acta Diabetol. 2012 Dec;49 Suppl 1:S253-7. doi: 10.1007/s00592-012-0433-y. Epub 2012 Oct 2. PMID 23053880
- [Background] Coggins M, Lindner J, Rattigan S, Jahn L, Fasy E, Kaul S, Barrett E. Physiologic hyperinsulinemia enhances human skeletal muscle perfusion by capillary recruitment. Diabetes. 2001 Dec;50(12):2682-90. doi: 10.2337/diabetes.50.12.2682. PMID 11723050
- [Background] Vincent MA, Clerk LH, Lindner JR, Price WJ, Jahn LA, Leong-Poi H, Barrett EJ. Mixed meal and light exercise each recruit muscle capillaries in healthy humans. Am J Physiol Endocrinol Metab. 2006 Jun;290(6):E1191-7. doi: 10.1152/ajpendo.00497.2005. PMID 16682488
- [Background] Zhang L, Vincent MA, Richards SM, Clerk LH, Rattigan S, Clark MG, Barrett EJ. Insulin sensitivity of muscle capillary recruitment in vivo. Diabetes. 2004 Feb;53(2):447-53. doi: 10.2337/diabetes.53.2.447. PMID 14747297
- [Background] Vincent MA, Dawson D, Clark AD, Lindner JR, Rattigan S, Clark MG, Barrett EJ. Skeletal muscle microvascular recruitment by physiological hyperinsulinemia precedes increases in total blood flow. Diabetes. 2002 Jan;51(1):42-8. doi: 10.2337/diabetes.51.1.42. PMID 11756321
- [Background] Vincent MA, Clerk LH, Lindner JR, Klibanov AL, Clark MG, Rattigan S, Barrett EJ. Microvascular recruitment is an early insulin effect that regulates skeletal muscle glucose uptake in vivo. Diabetes. 2004 Jun;53(6):1418-23. doi: 10.2337/diabetes.53.6.1418. PMID 15161743
- [Background] Inyard AC, Clerk LH, Vincent MA, Barrett EJ. Contraction stimulates nitric oxide independent microvascular recruitment and increases muscle insulin uptake. Diabetes. 2007 Sep;56(9):2194-200. doi: 10.2337/db07-0020. Epub 2007 Jun 11. PMID 17563063
- [Background] Clerk LH, Vincent MA, Barrett EJ, Lankford MF, Lindner JR. Skeletal muscle capillary responses to insulin are abnormal in late-stage diabetes and are restored by angiotensin-converting enzyme inhibition. Am J Physiol Endocrinol Metab. 2007 Dec;293(6):E1804-9. doi: 10.1152/ajpendo.00498.2007. Epub 2007 Oct 2. PMID 17911341
- [Background] Scognamiglio R, Negut C, De Kreutzenberg SV, Tiengo A, Avogaro A. Postprandial myocardial perfusion in healthy subjects and in type 2 diabetic patients. Circulation. 2005 Jul 12;112(2):179-84. doi: 10.1161/CIRCULATIONAHA.104.495127. Epub 2005 Jul 5. PMID 15998667
- [Background] Chai W, Liu J, Jahn LA, Fowler DE, Barrett EJ, Liu Z. Salsalate attenuates free fatty acid-induced microvascular and metabolic insulin resistance in humans. Diabetes Care. 2011 Jul;34(7):1634-8. doi: 10.2337/dc10-2345. Epub 2011 May 26. PMID 21617098
- [Background] Chan A, Barrett EJ, Anderson SM, Kovatchev BP, Breton MD. Muscle microvascular recruitment predicts insulin sensitivity in middle-aged patients with type 1 diabetes mellitus. Diabetologia. 2012 Mar;55(3):729-36. doi: 10.1007/s00125-011-2402-3. Epub 2011 Dec 14. PMID 22167126
- [Background] Westerbacka J, Uosukainen A, Makimattila S, Schlenzka A, Yki-Jarvinen H. Insulin-induced decrease in large artery stiffness is impaired in uncomplicated type 1 diabetes mellitus. Hypertension. 2000 May;35(5):1043-8. doi: 10.1161/01.hyp.35.5.1043. PMID 10818062
- [Background] Llaurado G, Ceperuelo-Mallafre V, Vilardell C, Simo R, Freixenet N, Vendrell J, Gonzalez-Clemente JM. Arterial stiffness is increased in patients with type 1 diabetes without cardiovascular disease: a potential role of low-grade inflammation. Diabetes Care. 2012 May;35(5):1083-9. doi: 10.2337/dc11-1475. Epub 2012 Feb 22. PMID 22357186
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Asmar R, Benetos A, Topouchian J, Laurent P, Pannier B, Brisac AM, Target R, Levy BI. Assessment of arterial distensibility by automatic pulse wave velocity measurement. Validation and clinical application studies. Hypertension. 1995 Sep;26(3):485-90. doi: 10.1161/01.hyp.26.3.485. PMID 7649586
- [Background] Baron AD. Hemodynamic actions of insulin. Am J Physiol. 1994 Aug;267(2 Pt 1):E187-202. doi: 10.1152/ajpendo.1994.267.2.E187. PMID 8074198